CLINICAL TRIAL: NCT04260152
Title: A Prospective, Randomized, Controlled, Double-blind, Multi-center Study to Assess Non-inferiority of Geistlich Fibro-Gide® in Comparison to Connective Tissue Graft for the Treatment of Recession Defects
Brief Title: Evaluation of Geistlich Fibro-Gide® + CAF in Comparison to CTG + CAF for the Treatment of Recession Defects at 6 Months
Acronym: GFG-US-REC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Collaborators: Medelis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10808-121
Record Dates: First submitted 2019-09-18; First posted 2020-02-07 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2020-03

CONDITIONS: Gingival Recession
Keywords: Gingival Recession; Fibro-Gide; CAF; CTG; Geistlich
MeSH Terms: conditions — Gingival Recession | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Split-mouth, randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind (Outcomes Examiner, Subject)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control: CAF + CTG (Active Comparator): Following root preparation and conditioning, the CTG is obtained from the palate according to the randomization scheme and shaped to the recipient site and may be sutured to the papilla region and the coronally advanced flap (CAF) is sutured into place.
  Interventions: Procedure: Connective Tissue Graft (CTG
- Test: CAF + Geistlich Fibro-Gide® (test) (Experimental): Following root preparation and conditioning, Geistlich Fibro-Gide® is cut to size and shaped to the recipient and may be sutured and the coronally advanced flap (CAF) is sutured into place.
  Interventions: Device: Geistlich Fibro-Gide

INTERVENTIONS:
Device: Geistlich Fibro-Gide — Surgical recession root coverage with coronally advanced flap in combination with Geistlich Fibro-Gide
  Other Names: Coronally advanced Flap (surgery/ procedure)
  Arms: Test: CAF + Geistlich Fibro-Gide® (test)
Procedure: Connective Tissue Graft (CTG — Surgical recession root coverage with coronally advanced flap in combination with CTG
  Other Names: Coronally advanced Flap (surgery/ procedure)
  Arms: Control: CAF + CTG

SUMMARY:
This double blind, randomized, split mouth study evaluates the non-inferiority of Geistlich Fibro-Gide® in comparison to connective tissue graft for the treatment of Miller Class I or II recession defects at 6 months post treatment.

DETAILED DESCRIPTION:
This double blind, randomized, split mouth study evaluates the non-inferiority of Geistlich Fibro-Gide® in comparison to connective tissue graft for the treatment of Miller Class I or II recession defects at 6 months post treatment.

A total sample size of 30 subjects (n=30) will be evaluated at 3 centers with 4 investigators. Power analysis based on 80% power and past McGuire/ Scheyer matched-pair defect recession coverage studies, with one-sided confidence interval 0.025, indicates that in order to detect a 12% difference in root coverage with ± 15% standard deviation a patient sample of 25 should be used . Given the multi-center nature of this study and the intention to follow patients long-term, with normal attrition, 30 subjects will ensure adequate long-term follow-up and provide a "power buffer" for any outcome differences that might be seen between centers.

30 Patients with Miller Class I or II recession defects on bilateral sites will be treated randomly with coronally advanced flap (CAF) in combination with either Geistlich Fibro-Gide (GFG =Test) on one side, and Connective Tissue Graft (CTG = Control) on the contralateral side of the mouth. Follow-up visits after visit 2 surgery will be conducted at week 1,2, 4,12 and 24 and in the long term after 1,3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age, inclusive.
* Subjects must have at least two teeth with buccal Miller Class I or II recession type defects, 3 mm deep and 3 mm wide on the same tooth in the contralateral quadrant of the same jaw
* Defects should be similar in size and morphology
* Teeth with root canals should be asymptomatic, completed at least 6 months prior
* At least 1mm KT
* Subjects with parafunctional habits must wear a bite guard to be included.

Exclusion Criteria:

* Participation within the previous 30 days in other investigational clinical trials.
* Class V restorations or abfractions that obliterate the CEJ.
* Subjects whose teeth have extremely prominent root surfaces -greater than 2mm facially to the adjacent teeth measured at the level of the CEJ.
* Systemic conditions that could influence wound healing or any other conditions that would preclude periodontal surgery.
* Taking medications that compromise wound healing.
* Acute infectious lesions in the areas intended for surgery.
* Untreated moderate to severe periodontal disease.
* Weekly or more frequent use of nicotine products within the past 6 months.
* Females who are pregnant or lactating, or sexually active female subjects who are of childbearing potential and who are not using hormonal or barrier methods of birth control.
* Subjects who require sedation in order to undergo surgery.
* Molars, teeth with axial mobility or interproximal loss of attachment, or full coverage crowns or veneers do not qualify.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Change in percent root coverage | 6 months post-treatment
  Change in percent root coverage compared to baseline

SECONDARY OUTCOMES:
Safety Endpoints: number and frequency of (S)AEs over all and by organ class | 1, 2, 4, 7, 12 and 24 weeks and year 1,3 and 5 post treatment
  Assessment of (S)AEs starting at Visit 2, Surgery
General Periodontal Examination (GPE) | baseline (day 0) and 6 months; 1, 3, 5 years post-treatment
  change of GPE at various visits compared to baseline, scoring codes 0-4
Assessment of Wound Healing | 1, 2, 4, 12 weeks post-treatment
  Judgement of soft tissue wound healing after surgery at Visits 3-6; Primary complete wound closure? yes = complete/ no = dehiscence visible
Assessment of Wound Healing | 1, 2, 4, 12 weeks post-treatment
  Judgement of soft tissue wound healing after surgery at Visits 3-6; if dehiscence visible, dehiscence size: lenght and width in mm
Assessment of Wound Healing | 1, 2, 4, 12 weeks post-treatment
  Judgement of soft tissue wound healing after surgery at Visits 3-6; presence of Swelling (yes/ no),
Overall Duration of Treatment Surgery | 2-6 hours at day of surgery
  Interval from surgery start until surgery end in Hours/Minutes
Patient Reported Outcome (PRO) -Patient Diary: Discomfort | 7 days after surgery starting 1 day after surgery
  Post-Op PRO Discomfort Diary completed by Patients at home; scale 0-10, 0=no pain or discomfort at all, 10=as much as you can imagine,
Patient Reported Outcome (PRO) -Questionnaire: Esthetics | 6 months, 1, 3, 5 years post-treatment
  Post-Op PRO questionnaire, Esthetics and overall satisfaction, patients will be asked by a 3rd party recorder, scale 0-10, 0=not satisfied at all with estehtic appearance, 10=completely satisfied,
Patient Reported Outcome (PRO) -Questionnaire: for surgical preference | 1, 2, 4, 12 weeks, 6 months, 1, 3, 5 years post-treatment
  Post-Op PRO questionnaire, Surgival procedure Preference, patients will be asked by a 3rd party recorder, Overall which treatment did you prefer? A or B
Safety endpoints: Concomitant Medication | 1, 2, 4, 12 weeks, 6 months, 1, 3, 5 years post-treatment
  Use of Concomitant medication Review: Type of concomitant Medication used.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K McGuire, DDS MSD, Principal Investigator — PerioHealth Professionals
Locations (3):
- United States (3):
  - Seven Lakes Periodontitis, Fenton, Michigan
  - Perio Health Professionals, Houston, Texas
  - Oral Health Specialists, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No